CLINICAL TRIAL: NCT05143840
Title: Asciminib as Initial Therapy With Addition of Lower Dose Tyrosine Kinase Inhibitors for Patients With Chronic Myeloid Leukemia Who do Not Achieve Optimal Response or a Deep Molecular Remission (ALERT CML)
Brief Title: Asciminib as Initial Therapy for Patients With Chronic Myeloid Leukemia in Chronic Phase
Acronym: ALERTCML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: H. Jean Khoury Cure CML Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HJKC3-0004; CABL001AUS06T (Other: Novartis Study Identifier)
Record Dates: First submitted 2021-11-16; First posted 2021-12-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-02

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase; Adult CML; Leukemia, Myeloid; Leukemia,Myeloid, Chronic
Keywords: Chronic Myeloid Leukemia; Adult CML; tyrosine kinase inhibitors; H. Jean Khoury Cure CML Consortium; HJKC3-0004
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — asciminib

STUDY DESIGN:
Intervention Model Description: Single group frontline asciminib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single Agent Asciminib Arm (Experimental): Asciminib 80mg Asciminib will be taken orally once a day starting cycle 1 day 1 for up to 24 months during the single agent asciminib phase.
  Patients will receive asciminib orally 80mg orally once a day starting cycle 1 day 1 for up to 24 months during the single agent asciminib phase.
  Interventions: Drug: Single Agent Asciminib
- Adding Low TKI (Experimental): TKI should begin within 28-days of obtaining central eligibility confirmation. This phase II trial will use single agent asciminib 80 mg PO daily during the single agent asciminib phase. All eligible subjects will begin asciminib on cycle 1 day 1 of this trial.
  Low dose tyrosine kinase inhibitor (lowTKI) (dasatinib 50 mg daily or imatinib 300 mg daily or nilotinib 300 mg daily) at investigators discretion, may be added to asciminib in the following situations:
  * Patients who have treatment failure at any time based on ELN criteria (Appendix 7)
  * Patients who have a warning response after 12 months of single agent asciminib based on ELN criteria (Appendix 7)
  * Patients who have not achieved MR4.5 after 24 months, but no later than 36 months, of single agent asciminib.
  Interventions: Combination Product: Low TKI
- Elective treatment free remission arm: (Experimental): .Elective treatment free remission arm: Once central eligibility has been obtained the patient should discontinue asciminib and if applicable lowTKI within 14 days.
  Interventions: Other: Elective Free Treatment

INTERVENTIONS:
Drug: Single Agent Asciminib — taken orally once a day starting cycle 1 day 1 for up to 24 months during the single agent asciminib phase. Asciminib is a potent allosteric inhibitor of BCR::ABL1.
  Other Names: ABL001
  Arms: Single Agent Asciminib Arm
Combination Product: Low TKI — Low dose tyrosine kinase inhibitor (lowTKI) (dasatinib 50 mg daily or imatinib 300 mg daily or nilotinib 300 mg daily) at investigators discretion, may be added to asciminib in the following situations:
  * Patients who have treatment failure at any time based on ELN criteria (Appendix 7)
  * Patients who have a warning response after 12 months of single agent asciminib based on ELN criteria (Appendix 7)
  * Patients who have not achieved MR4.5 after 24 months, but no later than 36 months, of single agent asciminib.
  Arms: Adding Low TKI
Other: Elective Free Treatment — Once central eligibility has been obtained the patient should discontinue asciminib and if applicable lowTKI within 14 days.
  Arms: Elective treatment free remission arm:

SUMMARY:
This study is a multicenter Phase 2, non-randomized, open-label single-group frontline study administering asciminib in patients with newly diagnosed Chronic Myeloid Leukemia-Chronic Phase (CML-CP). The aim of this study is to evaluate the efficacy and safety of asciminib in newly diagnosed CML-CP. Patients will receive asciminib 80 mg orally once daily during the single asciminib phase. Response is determined by PCR (polymerase chain reaction) blood test during the study. Patients who have not achieved a response after 24 months (but no later than 36 months) of single agent asciminib will be offered the addition of a low dose tyrosine kinase inhibitor (low-TKI) namely dasatinib, imatinib, or nilotinib at the investigator's discretion. The following doses of the TKIs will be used:

1. Dasatinib 50 mg daily
2. Imatinib 300 mg daily
3. Nilotinib 300 mg daily

Patients will discontinue study treatment if they experience disease progression, or unacceptable toxicity.

DETAILED DESCRIPTION:
Asciminib is a potent allosteric inhibitor of BCR-ABL1 oncogene that confers resistance to tyrosine kinase inhibitors (TKIs). Asciminib has potential to combine with TKIs to prevent the emergence of BCR-ABL1 mutations, increasing the depth of molecular response in CML-CP patients. Anticipated enrollment is 50 subjects across sites.

Primary Objective:

To estimate the proportion of patients with previously untreated CML-CP who attain BCR::ABL1 <0.01% (MR4.0) IS by RQ-PCR with single agent asciminib therapy.

Secondary Objectives:

1. To estimate the proportion of patients achieving molecular response at specific time points
2. To estimate the time to molecular response
3. To evaluate the duration of hematologic and molecular response to asciminib
4. To define the time to progression and overall survival for patients with CML in early CP treated with asciminib
5. To evaluate the safety profile of asciminib in patients with CML-CP
6. To evaluate the development of ABL mutations for patients with CML in early CP treated with asciminib
7. To analyze differences in response rates and in prognosis within different risk groups and patient characteristics
8. To evaluate patient-reported outcomes in patients with CML receiving asciminib
9. To investigate treatment-free remission after at least 2 years of sustained deep molecular remission for patients receiving single agent asciminib or combination (asciminib + low TKI)

Exploratory objectives:

1. To evaluate the safety and efficacy of concomitant use of low TKI with asciminib in patients who have not achieved MR4.5.
2. To evaluate the rate of successful treatment discontinuation for patients using the combination of asciminib and low TKI
3. To evaluate the safety and efficacy of concomitant use of lowTKI with asciminib in patients who experience treatment failure at any time with single agent asciminib
4. To evaluate the safety and efficacy of concomitant use of lowTKI with asciminib in patients who have not achieved an optimal response after 12 months of single agent asciminib
5. Evaluate the role of Digital droplet PCR (ddPCR) in predicting TFR
6. Evaluating the correlation between the gene expression signature of patients and the chances of achieving MMR and DMR
7. Evaluate whether B, NK and T cells DNA mutation and RNA expression are relevant and whether they can predict response in patients with CML using single cell analysis.

Subjects must meet all inclusion criteria and none of the exclusion criteria of the study. No enrollment waivers will be granted. After successful screening, subjects will be enrolled and treatment will start within 7 days of enrollment. Eligible subjects will begin asciminib on cycle 1 day 1 of the trial. After 2 years (but no later than 3 years), subjects will be offered the addition of taking nilotinib, dasatinib, or imatinib with asciminib if a molecular response is not met (PCR blood test).

Duration of each participant is expected to take approximately 5 years on treatment and up to a total of 8 years if attempting treatment free remission.

Regimen Description

Asciminib 80 mg Oral Once a day 4 weeks (28 days) Nilotinib 300 mg* Oral Once a day 4 weeks (28 days) Dasatinib 50 mg* Oral Once a day 4 weeks (28 days) Imatinib 300 mg* Oral Once a day 4 weeks (28 days)

*Nilotinib, dasatinib, or imatinib will be taken if indicated.

Dose levels and dose modifications of the study drugs will be made per protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Willing and able to give informed consent
3. Newly diagnosed with CML in chronic phase within 6 months from confirmed diagnosis via bone marrow biopsy/aspirate and have either the b3a2 (e14a2) or b2a2 (e13a2) variants that give rise to the p210 BCR::ABL1 protein. Subtype classification whether b3a2 (e14a2) or b2a2 (e13a2) is not required for study eligibility.
4. Minimal prior CML therapy with a TKI for less than or equal to 30 days. Treatment with hydroxyurea, busulfan, anagrelide or other non-specific chemotherapy agents is allowed with no time restrictions within the eligible time from diagnosis.
5. ECOG performance status 0-2 (appendix 1)
6. Adequate organ function:

   * AST and ALT < 3 times the institutional upper limit of normal (ULN)
   * eGFR ≥ 30 mL/min as calculated using the 2021 chronic kidney disease epidemiology (CKD-EPI) creatinine equation (https://www.kidney.org/professionals/kdoqi/gfr_calculator)
   * Total bilirubin < 1.5 times the institutional ULN or < 3.0 x the institutional ULN with Gilbert Syndrome (unless direct bilirubin is within normal limits)
7. Adequately controlled blood pressure, defined as systolic blood pressure of <140 mmHq and diastolic of <90 mmHg, at the time of enrollment.
8. Lipase ≤ 1.5 x ULN. For lipase > ULN - ≤ 1.5 x ULN, value should be considered not clinically significant and not associated with risk factors for acute pancreatitis.
9. Creatine phosphokinase < 2.5 x ULN
10. Female patients must meet one of the following:

    1. Postmenopausal for at least one year before the screening visit,
    2. Surgically sterile
    3. If they are of childbearing potential, agree to practice two effective methods of contraception from the time of signing of the informed consent form through 90 days after the last dose of study drug,
    4. Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable
    5. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)
11. Male patients, even if surgically sterilized (i.e., status post vasectomy), must agree to one of the following:

    1. Practice effective barrier contraception during the entire study treatment period and through 90 days after the last study drug dose
    2. Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable
    3. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

1. Patients with accelerated or blast phase CML (refer to appendix 4)
2. Active second malignancy requiring active treatment
3. History of recent (within 12 months) acute pancreatitis or chronic pancreatitis
4. Subjects who have previously received treatment with asciminib.
5. Subjects with PLT count < 50,000 mm3 or ANC of < 500 mm3 or Hemoglobin < 8 g/dL
6. Cardiac or cardiac repolarization abnormality, including any of the following:

   1. History within 6 months prior to starting study treatment of myocardial infarction (MI), angina pectoris, coronary artery bypass graft (CABG)
   2. Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third degree AV block)
   3. QTcF at screening greater than or equal to 450 msec (male patients), greater than or equal to 460 msec (female patients) unless patient has a pacemaker
   4. Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

   i. Risk factors for Torsades de Pointes (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia ii. Concomitant medication(s) with a "Known risk of Torsades de Pointes" per wwwcrediblemeds.org/ that cannot be discontinued or replace 7 days prior to starting study drug by safe alternative medication.

   iii. Inability to determine the QTcF interval
7. Pregnant or lactating
8. Taking a strong inhibitors or inducers of CYP3A4 or CYP3A4 substrates with narrow therapeutic index (refer to appendix 6) at time of enrollment
9. Unable to comply with lab appointment schedule and PRO assessments
10. Another investigational drug within 4 weeks of enrollment
11. Any serious medical or psychiatric illness that could, in the investigator's opinion, interfere with the completion of treatment according to this protocol
12. Patient has undergone a prior allogeneic stem cell transplant
13. Known clinical history of active HBV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2032-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure 1: Deep Molecular Response | 24 months
  The proportion of patients achieving BCR::ABL1 <0.01% IS (MR4.0) within 12 months of treatment with single agent asciminib
Digital Droplet PCR | 2 years
  Digital droplet PCR (ddPCR). Our Consortium work in the LAST study showed that ddPCR is more sensitive than conventional PCR and is very important in predicting TFR in detecting BCR::ABL1 in cases without detectable disease by conventional PCR29. Thus, samples taken for BCR::ABL1 monitoring in this trial will also be tested by ddPCR using the Bio-Rad platform. This will allow for a head to head comparison of these two methods.

SECONDARY OUTCOMES:
The rates of BCR::ABL1 IS ≤10%, ≤1% (MR2), ≤0.1% (MMR), ≤0.01% (MR4), and ≤0.0032% MR4.5 | 2 years
  The rates of BCR::ABL1 IS ≤10%, ≤1% (MR2), ≤0.1% (MMR), ≤0.01% (MR4), and ≤0.0032% MR4.5 by 3, 6, 12, 18, and 24 months of therapy
Time to complete hematological response. | 2 years
  Time to complete hematological response (CHR), MR1, MR2, MMR, MR4.0, MR4.5
Duration of MR1, MR2, MMR, MR4.0, MR4.5, and undetectable BCR::ABL1. | 2 years
  Duration of MR1, MR2, MMR, MR4.0, MR4.5, and undetectable BCR::ABL1.
FFS, TFS, EFS, and OS | 2 years
  4. Failure-free (FFS), transformation-free (TFS), event-free (EFS), and overall (OS) survival.
Adverse Events | 2 years
  The rates of adverse events related to asciminib
ABL1 sequencing at the time of primary resistance | 2 years
  ABL1 sequencing at the time of primary resistance and test the diagnostic sample for the specific ABL mutation found at resistance (if any).
Clonal evolution and Sokal risk score | 2 years
  Evaluate response and clinical outcomes by presence of clonal evolution, or Sokal risk score at diagnosis.
Patient Reported Outcomes | 2 years
  Patient-reported outcomes at various timepoints per schedule of events.
Rate of MMR loss | 2 years
  Evaluate the rate of MMR loss after asciminib discontinuation for an attempt at treatment free remission at 6 and 24 months from stopping therapy.

OTHER OUTCOMES:
Adverse Events when low TKI added | 2 years
  The rates of adverse events with asciminib + low dose TKI
Loss of MMR | 2 years
  Evaluate rate of loss of MMR after treatment discontinuation for patients reaching sustained MR4.5 with asciminib and lowTKI 6 and 24 months from stopping therapy
Evaluate the rates of BCR::ABL1 | 2 years
  Evaluate the rates of BCR::ABL1 IS ≤10% (MR1), ≤1% (MR2), ≤0.1% (MMR), ≤0.01% (MR4), and ≤0.0032% (MR4.5) by 3, 6, 12, 18, and 24 months of combination therapy for patients who experience treatment failure at any time with asciminib alone
Rate of MR4.5 after addition of low TKI | 2 years
  Evaluate the rate of MR4.5 by 6 and 12 months after addition of lowTKI for patients not in MR4.5 after 24 months of asciminib alone.
rates of BCR::ABL1 for patients who have a warning response after 12 months of asciminib | 2 years
  Evaluate the rates of BCR::ABL1 IS ≤10% (MR1), ≤1% (MR2), ≤0.1% (MMR), ≤0.01% (MR4), and ≤0.0032% (MR4.5) by 3, 6, 12, 18, and 24 months of combination therapy for patients who have a warning response after 12 months of asciminib alone
Loss of MMR after treatment discontinuation | 2 years
  Evaluate rate of loss of MMR after treatment discontinuation for patients reaching sustained MR4.5 with asciminib and lowTKI 6 and 24 months from stopping therapy
Gene expression signature | 2 years
  Gene expression signature. Recently completed work by the Radich Lab with Novartis revealed a signature of response in patients treated on the ENESTnd trial31. Most of the genes and pathways associated with MMR and DMR involved upregulation of immune pathways. We will test if similar phenomenon is occurring with asciminib response by performing RNAseq on all pre-treatment trials. Analysis of the data will be performed in the same manner as the ENESTnd biomarker study.
Single cell analyses | 2 years
  Single cell analyses. As noted above, response to nilotinib and imatinib appear to involve the immune system. However, at diagnosis these cells (B, NK, T) are not plentiful. What cells are driving this response? We will use the "tri-omics" platform from Mission Biosciences to sort single cells by cell type, and then perform DNA mutational analyses (myeloid leukemia genes) and RNA expression. This will allow us to determine how many cells of each type are present, whether they have other relevant mutations, and if they are responsible for the immune signal.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — Augusta University
Locations (7):
- United States (7):
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin